CLINICAL TRIAL: NCT04564040
Title: A 2-Part, Phase I, Open-label, Single-dose, Sequential, Randomized, Crossover Study of Acalabrutinib Tablet Suspension Delivered Via Nasogastric Tube in Healthy Subjects to Evaluate Relative Bioavailability and Proton-pump Inhibitor (Rabeprazole) Effect
Brief Title: A Study in Healthy Subjects to Assess Bioavailability (Proportion of a Drug Which Enters the Circulation to Have an Active Effect) of Acalabrutinib Tablet and Protonpump Inhibitor Effect (Members of a Class of Medications That Inhibits in Gastric Acid Production) for Rabeprazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D8223C00005
Record Dates: First submitted 2020-08-27; First posted 2020-09-25 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Mantle Cell Lymphoma; COVID-19
Keywords: Sequential; Proton-pump Inhibitor; Relative Bioavailability; Bruton Tyrosine Kinase Inhibitor
MeSH Terms: conditions — Lymphoma, Mantle-Cell; COVID-19 | interventions — acalabrutinib; Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Acalabrutinib Treatment Sequence 1 (Experimental): Part 1: Participants will receive Treatment A (100 mg AT suspension in water via NG administration) in Period 1, Treatment B (100 mg acalabrutinib capsule suspension via NG administration) in Period 2, and Treatment C (100 mg AT suspension in water via NG administration plus 20 mg rabeprazole) in Period 3.
  Part 2: Participants will receive Treatment D (100 mg AT suspension in water via NG administration) in Period 1 and Treatment A in Period 2.
  Interventions: Drug: Acalabrutinib Treatment A; Drug: Acalabrutinib Treatment B; Drug: Acalabrutinib Treatment C; Drug: Acalabrutinib Treatment D
- Acalabrutinib Treatment Sequence 2 (Experimental): Part 1: Participants will receive Treatment B in Period 1, Treatment A in Period 2, and Treatment C in Period 3.
  Part 2: Participants will receive Treatment A in Period 1 and Treatment D in Period 2.
  Interventions: Drug: Acalabrutinib Treatment A; Drug: Acalabrutinib Treatment B; Drug: Acalabrutinib Treatment C; Drug: Acalabrutinib Treatment D

INTERVENTIONS:
Drug: Acalabrutinib Treatment A — Participants will receive 100 mg AT suspension in water via NG tube.
  Other Names: AT
Drug: Acalabrutinib Treatment B — Participants will receive 100 mg acalabrutinib capsule suspension via NG tube.
  Other Names: Acalabrutinib capsule
Drug: Acalabrutinib Treatment C — Participants will receive 100 mg AT suspension in water via NG administration plus 20 mg rabeprazole.
  Other Names: AT and Pariet® (raberprazole)
Drug: Acalabrutinib Treatment D — Participants will receive 100 mg AT orally.
  Other Names: AT

SUMMARY:
This Phase 1 study is being conducted to support the clinical development of acalabrutinib in hospitalized patients who are unable to swallow acalabrutinib tablet or capsule due to respiratory failure, eg, they may require endotracheal intubation for ventilator support and nasogastric (NG) tube placement, and it is important to have a clinically acceptable method to administer acalabrutinib via NG tube.

Part 1 of the study is designed to evaluate relative bioavailability by comparing the pharmacokinetic (PK) of AT suspension in water administered via NG tube with the PK of acalabrutinib capsule suspension in flat COCA-COLA administered via NG tube. Additionally, the PPI effect will be evaluated by comparing the PK of AT suspension in water administered via NG tube plus rabeprazole with the PK of AT suspension in water administered via NG tube.

Part 2 of the study is designed to evaluate the effect of NG administration on AT by comparing the PK of AT suspension in water administered via NG tube with the PK of AT orally administered with water.

DETAILED DESCRIPTION:
Part 1 of the study comprises:

* A screening period of maximum 28 days.
* Three treatment periods during which subjects will reside in the Clinical Unit from Day -2, Treatment Period 1 until at least 48 hours after dosing on Day 1, Treatment Period 3, ie, subjects will be discharged the morning of Day 3, Treatment Period 3.
* A Follow-up Visit within 7 to 10 days after the last dose of acalabrutinib.

There will be a minimum washout period of 4 days between treatment periods. Up to 20 subjects will be included to ensure at least 16 subjects are evaluable. Subjects will be randomized to one of 2 treatment sequences (ABC, BAC) and each subject will receive single doses of 3 treatments under fasted conditions.

Part 2 of the study comprises:

* A screening period of maximum 28 days.
* Two treatment periods during which subjects will reside in the Clinical Unit from Day -2, Treatment Period 1 until at least 48 hours after dosing on Day 1, Treatment Period 2, ie, subjects will be discharged the morning of Day 3, Treatment Period 2.
* A Follow-up Visit within 7 to 10 days after the last dose of acalabrutinib.

There will be a minimum washout period of 4 days between treatment periods. Up to 20 subjects will be included to ensure at least 16 subjects are evaluable. Subjects will be randomized to one of 2 treatment sequences (DA, AD) and each subject will receive single doses of 2 treatments under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent form (ICF) prior to any study-specific procedures.
* Healthy adult male and female subjects aged 18 to 55 years (inclusive) with suitable veins for cannulation or repeated venipuncture.
* Male subjects and their female partners/spouses must adhere to the contraception methods.
* Female subjects must have a negative pregnancy test at screening and on admission, must not be lactating, and must be of non childbearing potential, confirmed at screening.
* Have a body mass index between 18.5 and 30 kg/m^2, inclusive, and weigh at least 50 kg and no more than 100 kg, inclusive, at screening.
* Understands the study procedures in the ICF and willing and able to comply with the protocol.

Exclusion Criteria:

* History or presence of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
* History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs, as judged by the Investigator.
* Any clinically significant illness, medical/surgical procedure, or trauma within 30 days of the first administration of study medication.
* Any clinically significant abnormalities in hematology, coagulation, clinical chemistry, or urinalysis results, at screening and on first admission to the Clinical Unit, as judged by the Investigator and defined as:

  (i) Hemoglobin less than lower limit of normal. (ii) Platelet count less than lower limit of normal. (iii) Absolute neutrophil count less than the lower limit of normal. (iv) Prothrombin time, Activated partial thromboplastin time or International normalized ratio above upper limit of normal (ULN).

  (v) Serum alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP) or serum bilirubin (total and direct) > 1.5 ULN.
* Any clinically significant abnormal findings in vital signs at screening and on first admission to the Clinical Unit, as judged by the Investigator, eg:

  (i) Systolic blood pressure (BP) < 90 mmHg or ≥ 140 mmHg and diastolic blood pressure (DBP) < 50 mmHg or ≥ 90 mmHg sustained for at least 10 minutes while resting in a supine position.

(ii) Pulse < 50 beats per minute (bpm) or > 90 bpm.

* Any clinically significant abnormalities on standard 12-lead electrocardiogram (ECG) at screening and on first admission to the Clinical Unit, including but not limited to any of the following:

  (i) QTcF > 450 millisecond (ms) or < 340 ms or family history of long QT syndrome, (ii) Any significant arrhythmia, (iii) Conduction abnormalities: Clinically significant PR (PQ) interval prolongation (> 240 ms); intermittent second or third degree atrioventricular (AV) block, or AV dissociation, Complete bundle branch block and/or QRS duration > 120 ms.
* Any positive result on screening for serum hepatitis B virus antigen or hepatitis B core antibody, hepatitis C antibody, and human immunodeficiency virus antibody.
* Has received a new chemical or biological entity within 90 days or at least 5 half-lives, whichever is the longest, of the first administration of study medication in this study.
* Plasma donation within 30 days of screening or any blood donation/loss more than 500 mL during the 90 days prior to screening.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to acalabrutinib or rabeprazole.
* Current smokers or those who have smoked or used nicotine products (including e cigarettes) within the 90 days prior to screening.
* Positive screen for drugs of abuse or cotinine at screening and on each admission to the Clinical Unit; positive screen for alcohol on each admission to the Clinical Unit.
* Treatment with a strong CYP3A inhibitor (within 14 days before first administration of study medication) or strong CYP3A inducer (within 28 days before first administration of study medication).
* Use of any prescribed or non prescribed medication.
* Known or suspected history of alcohol or drug abuse, or excessive intake of alcohol as judged by the Investigator.
* Excessive intake of caffeine-containing drinks or food as judged by the Investigator.
* Involvement of any AstraZeneca, Acerta Pharma, Parexel or study site employee or their close relatives.
* Judgment by the Investigator that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
* Subjects who cannot communicate reliably with the Investigator.
* Vulnerable subjects, eg, kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.
* Inability to swallow ATs or have a NG tube placed on separate occasions.
* History of a disorder which would make NG tube placement contraindicated, eg, esophageal strictures, esophageal varices, or bleeding diathesis.
* Evidence of ongoing systemic bacterial, fungal, or viral infection.
* Subject has a positive test result for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) reverse transcriptase polymerase chain reaction before randomization.
* Subject has clinical signs and symptoms consistent with corona virus disease 2019 (COVID-19), eg, fever, dry cough, dyspnea, sore throat, fatigue, or confirmed infection by appropriate laboratory test within the last 4 weeks prior to screening or on admission.
* History of severe COVID-19 (hospitalization, extracorporeal membrane oxygenation, mechanically ventilated).
* Subjects who are regularly exposed to COVID-19 as part of their daily life.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
Part 1 and 2: Area under plasma concentration-time curve from time zero to infinity (AUCinf) | Day 1 (pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours post-dose), Day 2 (24 hours post-dose)
  Part 1: Comparison of AUCinf of acalabrutinib and its metabolite (ACP-5862) following NG administration of AT suspension versus NG administration of acalabrutinib capsule suspension and to evaluate the effect of PPI (rabeprazole) on acalabrutinib and ACP-5862 PK profiles following NG administration of AT suspension.
  Part 2: Comparison of AUCinf of acalabrutinib and ACP 5862 following NG administration of AT suspension versus oral administration of AT.
Part 1 and 2: Area under the plasma concentration time curve from time zero to time of last quantifiable concentration (AUClast) | Day 1 (pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours post-dose), Day 2 (24 hours post-dose)
  Part 1: Comparison of AUClast of acalabrutinib and its metabolite (ACP-5862) following NG administration of AT suspension versus NG administration of acalabrutinib capsule suspension and to evaluate the effect of PPI (rabeprazole) on acalabrutinib and ACP-5862 PK profiles following NG administration of AT suspension.
  Part 2: Comparison of AUClast of acalabrutinib and ACP 5862 following NG administration of AT suspension versus oral administration of AT.
Part 1 and Part 2: Maximum observed plasma concentration (Cmax) | Day 1 (pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours post-dose), Day 2 (24 hours post-dose)
  Part 1: Comparison of Cmax of acalabrutinib and its metabolite (ACP-5862) following NG administration of AT suspension versus NG administration of acalabrutinib capsule suspension and to evaluate the effect of PPI (rabeprazole) on acalabrutinib and ACP-5862 PK profiles following NG administration of AT suspension.
  Part 2: Comparison of Cmax of acalabrutinib and ACP 5862 following NG administration of AT suspension versus oral administration of AT.
Part 1 and Part 2: Area under the plasma concentration-time curve from time zero to 24 hours post dose (AUC0-24) | Day 1 (pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours post-dose), Day 2 (24 hours post-dose)
  Part 1: Comparison of AUC0-24 of acalabrutinib and its metabolite (ACP-5862) following NG administration of AT suspension versus NG administration of acalabrutinib capsule suspension and to evaluate the effect of PPI (rabeprazole) on acalabrutinib and ACP-5862 PK profiles following NG administration of AT suspension.
  Part 2: Comparison of AUC0-24 of acalabrutinib and ACP 5862 following NG administration of AT suspension versus oral administration of AT.
Part 1 and 2: Time to reach maximum observed plasma concentration (tmax) | Day 1 (pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours post-dose), Day 2 (24 hours post-dose)
  Part 1: Comparison of tmax of acalabrutinib and its metabolite (ACP-5862) following NG administration of AT suspension versus NG administration of acalabrutinib capsule suspension and to evaluate the effect of PPI (rabeprazole) on acalabrutinib and ACP-5862 PK profiles following NG administration of AT suspension.
  Part 2: Comparison of tmax of acalabrutinib and ACP 5862 following NG administration of AT suspension versus oral administration of AT.
Part 1 and 2: Half-life associated with terminal slope (λz) of a semi-logarithmic concentrationtime curve (t1/2) | Day 1 (pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours post-dose), Day 2 (24 hours post-dose)
  Part 1: Comparison of t1/2 of acalabrutinib and its metabolite (ACP-5862) following NG administration of AT suspension versus NG administration of acalabrutinib capsule suspension and to evaluate the effect of PPI (rabeprazole) on acalabrutinib and ACP-5862 PK profiles following NG administration of AT suspension.
  Part 2: Comparison of t1/2 of acalabrutinib and ACP 5862 following NG administration of AT suspension versus oral administration of AT.
Part 1 and 2: Mean residence time of the drug in the systemic circulation from zero to infinity (MRT) | Day 1 (pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours post-dose), Day 2 (24 hours post-dose)
  Part 1: Comparison of MRT of acalabrutinib and its metabolite (ACP-5862) following NG administration of AT suspension versus NG administration of acalabrutinib capsule suspension and to evaluate the effect of PPI (rabeprazole) on acalabrutinib and ACP-5862 PK profiles following NG administration of AT suspension.
  Part 2: Comparison of MRT of acalabrutinib and ACP 5862 following NG administration of AT suspension versus oral administration of AT.
Part 1 and 2: Terminal elimination rate constant (λz) | Day 1 (pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours post-dose), Day 2 (24 hours post-dose)
  Part 1: Comparison of λz of acalabrutinib and its metabolite (ACP-5862) following NG administration of AT suspension versus NG administration of acalabrutinib capsule suspension and to evaluate the effect of PPI (rabeprazole) on acalabrutinib and ACP-5862 PK profiles following NG administration of AT suspension.
  Part 2: Comparison of λz of acalabrutinib and ACP 5862 following NG administration of AT suspension versus oral administration of AT.
Part 1 and 2: Apparent total body clearance of drug from plasms after extravascular administration (acalabrutinib only (CL/F) | Day 1 (pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours post-dose), Day 2 (24 hours post-dose)
  Part 1: Comparison of CL/F of acalabrutinib and its metabolite (ACP-5862) following NG administration of AT suspension versus NG administration of acalabrutinib capsule suspension and to evaluate the effect of PPI (rabeprazole) on acalabrutinib and ACP-5862 PK profiles following NG administration of AT suspension.
  Part 2: Comparison of CL/F of acalabrutinib and ACP 5862 following NG administration of AT suspension versus oral administration of AT.
Part 1 and 2: Apparent volume of distribution during the terminal phase after extravascular administration (acalabrutinib only) (Vz/F) | Day 1 (pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours post-dose), Day 2 (24 hours post-dose)
  Part 1: Comparison of Vz/F of acalabrutinib and its metabolite (ACP-5862) following NG administration of AT suspension versus NG administration of acalabrutinib capsule suspension and to evaluate the effect of PPI (rabeprazole) on acalabrutinib and ACP-5862 PK profiles following NG administration of AT suspension.
  Part 2: Comparison of Vz/F of acalabrutinib and ACP 5862 following NG administration of AT suspension versus oral administration of AT.
Part 1 and 2: Metabolite to parent ratio based on AUCinf and/or AUClast (M:P[AUC]) | Day 1 (pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours post-dose), Day 2 (24 hours post-dose)
  Part 1: Comparison of M:P[AUC] of acalabrutinib and its metabolite (ACP-5862) following NG administration of AT suspension versus NG administration of acalabrutinib capsule suspension and to evaluate the effect of PPI (rabeprazole) on acalabrutinib and ACP-5862 PK profiles following NG administration of AT suspension.
  Part 2: Comparison of M:P[AUC] of acalabrutinib and ACP 5862 following NG administration of AT suspension versus oral administration of AT.
Part 1 and 2: Metabolite to parent ratio based on Cmax (M:P[Cmax]) | Day 1 (pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours post-dose), Day 2 (24 hours post-dose)
  Part 1: Comparison of M:P[Cmax] of acalabrutinib and its metabolite (ACP-5862) following NG administration of AT suspension versus NG administration of acalabrutinib capsule suspension and to evaluate the effect of PPI (rabeprazole) on acalabrutinib and ACP-5862 PK profiles following NG administration of AT suspension.
  Part 2: Comparison of M:P[Cmax] of acalabrutinib and ACP 5862 following NG administration of AT suspension versus oral administration of AT.

SECONDARY OUTCOMES:
Number of subjects with serious and non-serious adverse events | From screening visit (Day -28) to Follow-up visit (7-10 days after last dose or early termination)
  Part 1: To evaluate the safety and tolerability of AT suspension administered via NG tube and to evaluate the safety and tolerability of AT suspension via NG tube when co-administered with rabeprazole.
  Part 2: To evaluate the safety and tolerability of AT, administered orally.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Rainard Fuhr, Principal Investigator — Parexel
Locations (1):
- Research Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from
  AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home